CLINICAL TRIAL: NCT01704794
Title: Antioxidant Effect of the Extract of Jobelyn (Sorghum Bicolor) on the Quality of Life of Patients With Sickle Cell Disease
Brief Title: Quality of Life Study for Sickle Cell Patients Treated With Jobelyn (Sorghum Bicolor Extract)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lagos State University (Other)
Responsible Party: Principal Investigator, Dr. A. O. Dosunmu, CONSULTANT IN THE DEPARTMENT OF HAEMATOLOGY & BLOOD TRANSFUSION, LASUTH, Lagos State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LASUTH/SCD01/2012
Record Dates: First submitted 2012-10-03; First posted 2012-10-11 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Other Sickle-cell Disorders With Crisis, Unspecified
Keywords: Sickle Cell Anemia; Quality of Life; Antioxidant; Anti inflammatory; Sorghum bicolor
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Folic Acid; Proguanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Folic Acid + Paludrine +Jobelyn (500mg) (Active Comparator): Folic acid 5mg given twice daily. Paludrine 50mg to 20mg daily. Jobelyn 500mg once daily.
  Interventions: Dietary Supplement: Folic Acid + Paludrine + Jobelyn (500mg)
- Folic Acid + Paludrine +Jobelyn (250mg.) (Active Comparator): Folic Acid 5mg daily Paludrine 20 - 40mg daily Jobelyn 250mg daily
  Interventions: Drug: Folic Acid + Paludrine + Jobelyn (250mg)
- Folic Acid + Paludrine + Jobelyn (2mg) (Active Comparator): Folic Acid 5mg daily Paludrine 20 - 40mg daily Jobelyn 2mg daily
  Interventions: Dietary Supplement: Folic Acid + Paludrine + Jobelyn (2mg)

INTERVENTIONS:
Dietary Supplement: Folic Acid + Paludrine + Jobelyn (500mg) — Combination of routine drugs + Jobelyn
  Other Names: Routine drugs; Sorghum bicolor extract (Jobelyn 500mg)
  Arms: Folic Acid + Paludrine +Jobelyn (500mg)
Drug: Folic Acid + Paludrine + Jobelyn (250mg) — Standard routine drugs for treatment of SCD with 250mg Jobelyn
  Other Names: Routine drugs; Sorghum bicolor extract (250mg)
  Arms: Folic Acid + Paludrine +Jobelyn (250mg.)
Dietary Supplement: Folic Acid + Paludrine + Jobelyn (2mg) — Combination of Paludrine + Folic Acid and Jobelyn 2mg (Sorghum bicolor extract)
  Other Names: Other Names: Routine drugs; Jobelyn (Sorghum bicolor extract)
  Arms: Folic Acid + Paludrine + Jobelyn (2mg)

SUMMARY:
The purpose of this study is to determine the antioxidant effect of prolonged use of sorghum bicolor (jobelyn) to increase the level of plasma superoxide dismutase and glutathione reductase in patients with sickle cell disease and to determine if there is any improvement in the quality of life of the patients.

DETAILED DESCRIPTION:
Jobelyn is an extract of sorghum bicolor that is popular in Nigeria as a herbal food supplement. This extract has been shown to have a high oxygen radical absorbance capacity (ORAC 37,622micro mole TE/g) compared to other botanical preparations 1. A second proven property is its anti inflammatory effect with a selective COX 2 inhibition 2. It has also been shown to correct anaemia induced in experimental rabbit by trypanosome brucei brucei 3.

Jobelyn is being consumed as a herbal nutritional supplement in many disorders including sickle cell disease in Nigeria without complaint in over 15 years. The toxicology profile is impressive with a wide therapeutic range.

Nigeria is one of the countries with the largest burden of sickle cell disease. It is a chronic genetic disorder that accounts for absenteeism at school and at work place. There is also a significant shortening of the life span of the affected patients. Sickle cell anaemia presents with recurrent bone pains and progressive organ damage that affects negatively the quality of life of the patients. Available measures that have been in use include use of hydroxyurea, chronic and acute red cell transfusion and haematopoietic stem cell transplantation. These have limitations in terms of adverse effects, cost and availability.

The pathogenesis involves intracellular precipitation of the mutant haemoglobin, rigidity of the cell, adhesion of cells to the endothelium. These cause recurrent tissue hypoxia and reperfusion which cause release of reactive oxygen series and agents of inflammation. The extract of sorghum is therefore expected to improve the quality of life of these patients.

Previous work done, have not investigated the long time effect of the extract on the quality of life of sickle cell patients. This study is therefore designed to compare the quality of life of patients on 500mg daily, 250mg daily and 2mg daily of jobelyn using adjusted standard tools. The secondary outcomes to study are changes in indicators of inflammation and systemic antioxidants in these patients. The study period is 12 months so that the period shall involve all the weather conditions in the region.

ELIGIBILITY:
Inclusion Criteria:

1. AGE : 14 To 40 years
2. SEX: Both sexes
3. Homozygous for the S gene (SS)

Exclusion Criteria:

1. Age below 14 years and above 40 years
2. Evidence of organ failure i.e heart failure, renal failure
3. No consent for study
4. Poor adherence to treatment and irregular visit to the clinic
5. Presence of chronic inflammation
6. Pregnancy

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
number of severe bone pain crises and hospital admissions in one year | 12 months
  Use of health related quality of life measures tool SF-36 and self reporting questionnaires

SECONDARY OUTCOMES:
Antioxidant and anti-inflammatory effect | 12 months
  Increase in glutathion reductase, Increase in superoxide dismutase, Reduction in C reactive protein, Reduction in lactate dehydrogenase and Liver enzymes tests

CONTACTS AND LOCATIONS:
Overall Officials: A O Dosunmu, M.D., Principal Investigator — Lagos State University
Locations (1):
- Lagos State University Teaching Hospital, Ikeja, Lagos, Nigeria

REFERENCES:
- [Background] Brohan M, Jerkovic V, Collin S. Potentiality of red sorghum for producing stilbenoid-enriched beers with high antioxidant activity. J Agric Food Chem. 2011 Apr 27;59(8):4088-94. doi: 10.1021/jf1047755. Epub 2011 Mar 7. PMID 21381750
- [Background] Geera B, Ojwang LO, Awika JM. New highly stable dimeric 3-deoxyanthocyanidin pigments from sorghum bicolor leaf sheath. J Food Sci. 2012 May;77(5):C566-72. doi: 10.1111/j.1750-3841.2012.02668.x. Epub 2012 Apr 10. PMID 22489620
- [Background] Kayode AP, Nout MJ, Linnemann AR, Hounhouigan JD, Berghofer E, Siebenhandl-Ehn S. Uncommonly high levels of 3-deoxyanthocyanidins and antioxidant capacity in the leaf sheaths of dye sorghum. J Agric Food Chem. 2011 Feb 23;59(4):1178-84. doi: 10.1021/jf103963t. Epub 2011 Jan 25. PMID 21322653
- [Background] Yang L, Browning JD, Awika JM. Sorghum 3-deoxyanthocyanins possess strong phase II enzyme inducer activity and cancer cell growth inhibition properties. J Agric Food Chem. 2009 Mar 11;57(5):1797-804. doi: 10.1021/jf8035066. PMID 19256554
- [Background] Shih CH, Siu SO, Ng R, Wong E, Chiu LC, Chu IK, Lo C. Quantitative analysis of anticancer 3-deoxyanthocyanidins in infected sorghum seedlings. J Agric Food Chem. 2007 Jan 24;55(2):254-9. doi: 10.1021/jf062516t. PMID 17227050
- [Background] Hunt DM, Emerson SU, Wagner RR. RNA- temperature-sensitive mutants of vesicular stomatitis virus: L-protein thermosensitivity accounts for transcriptase restriction of group I mutants. J Virol. 1976 May;18(2):596-603. doi: 10.1128/JVI.18.2.596-603.1976. PMID 178900
- [Background] Burdette A, Garner PL, Mayer EP, Hargrove JL, Hartle DK, Greenspan P. Anti-inflammatory activity of select sorghum (Sorghum bicolor) brans. J Med Food. 2010 Aug;13(4):879-87. doi: 10.1089/jmf.2009.0147. PMID 20673059
- [Background] Park JH, Darvin P, Lim EJ, Joung YH, Hong DY, Park EU, Park SH, Choi SK, Moon ES, Cho BW, Park KD, Lee HK, Kim MJ, Park DS, Chung IM, Yang YM. Hwanggeumchal sorghum induces cell cycle arrest, and suppresses tumor growth and metastasis through Jak2/STAT pathways in breast cancer xenografts. PLoS One. 2012;7(7):e40531. doi: 10.1371/journal.pone.0040531. Epub 2012 Jul 6. PMID 22792362
- [Background] Wu L, Huang Z, Qin P, Yao Y, Meng X, Zou J, Zhu K, Ren G. Chemical characterization of a procyanidin-rich extract from sorghum bran and its effect on oxidative stress and tumor inhibition in vivo. J Agric Food Chem. 2011 Aug 24;59(16):8609-15. doi: 10.1021/jf2015528. Epub 2011 Jul 29. PMID 21780844
- [Background] Awika JM, McDonough CM, Rooney LW. Decorticating sorghum to concentrate healthy phytochemicals. J Agric Food Chem. 2005 Aug 10;53(16):6230-4. doi: 10.1021/jf0510384. PMID 16076098
- [Background] Gee L, Abbott J, Conway SP, Etherington C, Webb AK. Validation of the SF-36 for the assessment of quality of life in adolescents and adults with cystic fibrosis. J Cyst Fibros. 2002 Sep;1(3):137-45. doi: 10.1016/s1569-1993(02)00079-6. PMID 15463820
- [Background] Okochi,V.I.,Okpuzor J, Okubena M.O., Awoyemi A.K. 2003 . The Influence of African Herbal Formula on the haematological parameters of trypanosome infected rats. African Journal of Biotechnology. 2 (9), 312-316.
- [Background] Erah P,O., Asonye C.C. Okhamafe A.O. 2003. Response of trypanosome brucei brucei induced anaemiato a commercialherbal preparation. African Journal of Biotechnology. 2,9, 307-311.
- [Background] Ogwumike OO. Hemopoietic effect of aqueous extract of the leaf sheath of Sorghum bicolor in albino rats. African Journal of Biomedical. Research. (2002): Vol 5; 69 - 71
- [Background] Oladiji AT, Jacob TO, Yakubu MT. Anti-anaemic potentials of aqueous extract of Sorghum bicolor (L.) moench stem bark in rats. J Ethnopharmacol. 2007 May 22;111(3):651-6. doi: 10.1016/j.jep.2007.01.013. Epub 2007 Jan 18. PMID 17306481
- [Background] Akande IS, Oseni AA, Biobaku OA. Effects of aqueous extract of Sorghum bicolor on hepatic, histological and haematological indices in rats. Journal of Cell and Animal Biology 4(9), 137-142, 2010.
- [Background] Nwinyi FC, Kwanashie HO. Evaluation of aqueous methanolic extract of Sorghum bicolor leaf base for antinociceptive and anti-inflammatory activities. African Journal of Biotechnology, 8 (18), 4642-4649, 2009.
- [Background] Eniojukan JF, Bolajoko AA. Toxicological Profiles of Commercial Herbal Preperation, Jobelyn. International Journal of Health Research, 2(4), 369-374, 2009.
- [Background] USDA Database for the Oxygen Radical Absorbance Capacity (ORAC) of Selected Foods, Release 2, U.S. Department of Agriculture, 2010.